CLINICAL TRIAL: NCT01215604
Title: Characterization of the Involvement of Translation Initiation Factors in the Immune Response to Acute Infection in the Elderly and Very Elderly
Brief Title: Involvement of Translation Initiation Factors in the Immune Response in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10156-2010CTIL
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Elderly Patient; Infection
Keywords: elderly patients; acute infection; translation initiation factors; eIF4E; eIF4G
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples of elderly patients diagnosed with acute infection will be collected at admittance to Meir hospital and on recovery (24-48 hours without fever and leukocytosis)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators propose that the translation initiation factors eIF4E and eIF4GI may be involved in resolution of acute inflammation (regardless of age). Furthermore, the investigators suggest that differences in translation initiation factors state of activation may contribute to inflammation. Finally, the investigators hypothesize that differences in translation initiation factors state of activation may underlie the immune compromised state of the very elderly affording additional explanation for the heightened morbidity from infection in this group.

In the current study the investigators aim to test these hypotheses by measuring the levels of eIF4E and eIF4G, their regulators, and targets in elderly (65-84yrs) and very elderly (85yrs<) patients hospitalized at Meir hospital for acute infection and after their recovery (detailed in study design).

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (65<)
* hospitalized for acute infection (fever 38c<, leukocytosis)

Exclusion Criteria:

* patients with dementia who can not sign informed consent of institutional Helsinki committee
* patient with active cancer with active chemotherapy treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patient aged >65 years admitted to internal medicine or geriatric departments due to acute infection with fever and leukocytosis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Heffez Ayzenfeld, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel